CLINICAL TRIAL: NCT07309627
Title: Effect of Virtual Reality-Based Rehabilitation on Balance, Pain, Kinesiophobia, Depression, and Quality of Life in Individuals With Lumbar Disc Herniation
Brief Title: VR Therapy Effects in Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: deniz 1
Record Dates: First submitted 2025-11-14; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Arm 1 - Control Group Arm Title: Control Group Arm Type: Active Comparator Description: Participants in this group will receive standard physiotherapy interventions commonly used for the management of lumbar disc herniation.
  Intervention Intervention Name: Conventional Physiotherapy Intervention Type: Behavioral Intervention Description: A traditional physiotherapy program including supervised stretching, strengthening, and mobility exercises tailored for individuals with lumbar disc herniation.
  Assigned Arm: Control Group
  Interventions: Other: Conventional Physiotherapy
- Experimental Group (Experimental): Arm 2 - Experimental Group Arm Title: Experimental Group Arm Type: Experimental Description: Participants in this group will receive a virtual reality-based exercise program designed to improve balance, reduce pain, decrease kinesiophobia, and enhance quality of life.
  Intervention Intervention Name: Virtual Reality Exercise Program Intervention Type: Behavioral Intervention Description: A structured virtual reality-based exercise protocol including balance, core-strengthening, mobility tasks, and functional training tailored for lumbar disc herniation.
  Assigned Arm: Experimental Group
  Interventions: Other: Conventional Physiotherapy; Other: VR

INTERVENTIONS:
Other: Conventional Physiotherapy — TENS, superficial and deep heat therapy, and interferential current + strengthening, stretching, and postural correction exercises Three times per week for six weeks, each session lasting 40 minutes,
  Other Names: Virtual Reality
Other: VR — The Virtual Reality (VR) group : conventional treatment in combination with a VR application (Balance System Assessment System and Active Video Games), (consisting of six different games at three difficulty levels (beginner, intermediate, advanced).
  Each game lasted for 2 minutes and was repeated twice. Over six weeks, both groups completed a total of 18 sessions (3 sessions per week)
  Arms: Experimental Group

SUMMARY:
This study aims to evaluate the effects of incorporating virtual reality (VR) therapy into routine physical therapy (RPT) on balance, pain, kinesiophobia, quality of life, and depression in individuals diagnosed with lumbar disc herniation (LDH).

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate the effects of adding virtual reality (VR) therapy to routine physical therapy (RPT) on balance, pain, kinesiophobia, quality of life, and depression in individuals with lumbar disc herniation (LDH).

Methods:

A total of 93 patients diagnosed with LDH will be randomly assigned into two groups: an intervention group (n=47) and a control group (n=46). Both groups will undergo a conventional physical therapy program consisting of transcutaneous electrical nerve stimulation (TENS), vacuum interference, heat application, and ultrasound therapy. In addition to the conventional program, the intervention group will receive VR-based therapy.

Participants will be assessed at baseline and at the end of the intervention period using the following outcome measures: balance assessed by the Nintendo Balance Board-based Balance System; activities of daily living assessed by the Oswestry Disability Index; back pain intensity assessed by the Visual Analog Scale; kinesiophobia assessed by the Tampa Kinesiophobia Scale; quality of life assessed by the Short Form-36 questionnaire; and depression assessed by the Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of lumbar disc herniation (LDH)
* Sedentary lifestyle
* Presence of low back pain for at least 3 months
* No participation in physiotherapy or structured rehabilitation programs within the previous 6 months

Exclusion Criteria:

Exclusion Criteria

* History of spinal surgery or spinal trauma
* Presence of vestibular disorders
* Presence of neurological diseases
* Presence of cardiopulmonary diseases
* Presence of other musculoskeletal disorders affecting participation
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | 8 weeks
  The ODI is a 10-item questionnaire developed to assess functional impairment in individuals with back pain. It evaluates changes in self-care, lifting, walking, sitting, standing, sleeping, social life, travel, and pain. Each item is scored from 0 to 5, with the total score ranging from 0 to 50. The total score is then multiplied by 2 and expressed as a percentage, with higher scores indicating greater disability
SF-36 Quality of Life Scale | 8 weeks
  The SF-36 assesses quality of life across eight domains: physical functioning, bodily pain, general health perception, vitality, mental health, social functioning, and physical and emotional roles. Its validity and reliability in Turkey were established by Pınar et al.
Tampa Kinesiophobia Scale (TSK) | 8 weeks
  The TSK is a 17-item self-report questionnaire using a 4-point Likert scale to assess fear of movement and/or reinjury. Total scores are calculated by reverse-scoring items 4, 8, 12, and 16, with possible scores ranging from 17 to 68. Scores of 37 or higher indicate a high level of kinesiophobia
Beck Depression Inventory (BDI) | 8 weeks
  The Beck Depression Inventory (BDI) is a 21-item self-report Likert-type scale used to determine the frequency of depressive symptoms. Items are scored from 0 to 3, and the scale's validity and reliability in Turkey were established by Ulusoy et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Üsküdar Üniversitesi, Umraniye, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arias LFG, Zhang Y, Tijssen M, Wilhelm E. Virtual Reality Supported Neck Stretching Exercises to Improve Cervical Range of Motion. Annu Int Conf IEEE Eng Med Biol Soc. 2025 Jul;2025:1-7. doi: 10.1109/EMBC58623.2025.11253550. PMID 41336211
- [Background] Yuenyongchaiwat K, Chitjamnogchai C, Sermsinsaithong N, Tavonudomgit W, Mahawong L, Buranapuntalug S, Songsorn P, Thanawattano C. Benefit of home-based virtual reality aerobic exercise combined with resistance training for reversing sarcopenia and reducing depression in community-dwelling older adults with sarcopenia: a randomized control trial. Arch Gerontol Geriatr. 2026 Mar;142:106108. doi: 10.1016/j.archger.2025.106108. Epub 2025 Nov 29. PMID 41338160
- [Background] Dutta A, Hatjipanagioti K, Newsham MA, Leyland L, Rickson L, Buchanan A, Farkhatdinov I, Twamley J, Das A. Extended Reality Biofeedback for Functional Upper Limb Weakness: Mixed Methods Usability Evaluation. JMIR XR Spat Comput. 2025 Jun 3;2:e68580. doi: 10.2196/68580. eCollection 2025. PMID 41340847